CLINICAL TRIAL: NCT02193841
Title: Simple Bone Cysts in Kids (SBoCK)
Brief Title: Simple Bone Cysts in Kids
Acronym: SBoCK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, James Wright, Orthopaedic Surgeon, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000042364
Record Dates: First submitted 2014-07-04; First posted 2014-07-18 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Bone Cyst
Keywords: Simple bone cyst; Unicameral bone cyst
MeSH Terms: conditions — Bone Cysts | interventions — Curettage; Punctures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C & P (Active Comparator): Curettage with puncture (C & P) will be performed alone
  Interventions: Procedure: Curettage with puncture (C & P); Device: Curette
- C & P with Vitoss (Active Comparator): A predetermined amount of Vitoss morsels will be injected following the curettage and puncture (C & P)
  Interventions: Procedure: Curettage with puncture (C & P); Device: Curette; Device: Vitoss morsels

INTERVENTIONS:
Procedure: Curettage with puncture (C & P) — A curette will be inserted to scrape the contents of the cyst (curettage) and a hole in the cyst wall will be made (puncture) near the bone marrow cavity
Device: Curette — A small surgical instrument with a rounded edge designed for scraping
Device: Vitoss morsels — A bone substitute intended for use as a filler for voids or gaps in bones
  Other Names: Tri-calcium phosphate bone graft substitute
  Arms: C & P with Vitoss

SUMMARY:
Simple bone cysts (SBCs) are cysts filled with fluid that occur most frequently in the long bones (arms or legs) of children. There are many ways to treat SBCs but it is unclear if one is better than another. The purpose of this research trial is to compare the effectiveness of two common treatments that are used by surgeons today.

DETAILED DESCRIPTION:
In general, few randomized clinical trials have been undertaken in paediatric orthopaedics, and only one to date has addressed the problem of simple bone cysts (SBCs). Also known as unicameral bone cysts, they are the commonest bone lesion in children. Despite general opinion, these cysts do not resolve at skeletal maturity.

Many forms of treatment have been recommended but none, including the popular methods of corticosteroid or bone marrow injections, have reliably eradicated SBC. Although the lesions are considered benign (non-cancerous), they cause pain, frequently interfere with function, dramatically restrict play activity, may re-fracture leading to growth arrest and/or deformity, and cause enormous anxiety for children and their families.

With a well-developed network of surgeons and researchers, we will provide evidence comparing the effectiveness of two treatment interventions for SBC. More specifically, our goals for this study are:

1. to compare the rate of radiographic healing between two standard treatments including curettage with puncture alone, and curettage with puncture followed by injection with Vitoss morsels;
2. to identify prognostic radiographic factors associated with simple bone cyst healing and fracture;
3. to determine the impact of simple bone cyst on children/family functioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed simple bone cyst in a long bone (ie. arm or leg) within last 3 months
* At least 3 weeks must have elapsed since last fracture
* At least 3 months must have elapsed since last cyst treatment
* Patients and/or their legal representatives willing to provide written informed consent (and assent, when appropriate)
* Patients with stabilizing implants in the bone where the cyst is located

Exclusion Criteria:

* Patients with bone disease (ie. osteogenesis imperfecta, cancer, osteoporosis, Paget's disease)
* Pregnant or breastfeeding female
* Patients with cysts crossing the growth plate (area where bone grows)

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-03; Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cyst healing | 2 years
  Healing will be graded according to a 4-point modified Neer's classification by radiologists

SECONDARY OUTCOMES:
Clinical measures (Cyst features) | 1 and 2 years
  Cyst features (ie. appearance, size) will be described or measured from X-rays taken annually after treatment
Functional measures (Questionnaire scores) | 1 and 2 years
  Function in participants will be evaluated using self-reported questionnaires for activity level, perception of illness, and pain annually after treatment

CONTACTS AND LOCATIONS:
Overall Officials: James G. Wright, Principal Investigator — The Hospital for Sick Children; Sevan Hopyan, Principal Investigator — The Hospital for Sick Children
Locations (25):
- United States (11):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Loma Linda University, Loma Linda, California
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The John Hopkins Hospital, Baltimore, Maryland
  - Hospital for Joint Diseases, New York, New York
  - Hospital for Special Surgery, New York, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
- The Royal Children's Hospital, Melbourne, Australia
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital at London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Shriners Hospital for Children - Canadian Unit, Montreal, Quebec
- United Kingdom (5):
  - Alder Hey Children's Hospital, Liverpool
  - Great Ormond Street Hospital for Children, London
  - Royal Manchester Children's Hospital, Manchester
  - Nuffield Orthopaedic Centre, Oxford
  - Sheffield Children's Hospital, Sheffield

REFERENCES:
- [Background] Wright JG, Yandow S, Donaldson S, Marley L; Simple Bone Cyst Trial Group. A randomized clinical trial comparing intralesional bone marrow and steroid injections for simple bone cysts. J Bone Joint Surg Am. 2008 Apr;90(4):722-30. doi: 10.2106/JBJS.G.00620. PMID 18381307
- [Background] Donaldson S, Wright JG. Recent developments in treatment for simple bone cysts. Curr Opin Pediatr. 2011 Feb;23(1):73-7. doi: 10.1097/MOP.0b013e3283421111. PMID 21191299
- [Background] Canavese F, Wright JG, Cole WG, Hopyan S. Unicameral bone cysts: comparison of percutaneous curettage, steroid, and autologous bone marrow injections. J Pediatr Orthop. 2011 Jan-Feb;31(1):50-5. doi: 10.1097/BPO.0b013e3181ff7510. PMID 21150732
- [Background] Donaldson S, Chundamala J, Yandow S, Wright JG. Treatment for unicameral bone cysts in long bones: an evidence based review. Orthop Rev (Pavia). 2010 Mar 20;2(1):e13. doi: 10.4081/or.2010.e13. PMID 21808696
- See also: SBoCK Trial Website — http://www.sickkids.ca/research/sbock/